CLINICAL TRIAL: NCT06902532
Title: Effectiveness of Coconut Oil Pulling With Clove Oil, Coconut Oil Pulling and Fluoride Mouthwash on Streptococcus Mutans Count in Children
Acronym: COPCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kholoud shaaban abdelmonaem mohamed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COPCO-2025; self funded study (Other: Cairo university-faculty of dentistry)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries
Keywords: Tooth Decay Streptococcus Mutans Oil Pulling Coconut Oil Clove Oil Fluoride Mouthwash Pediatric Dentistry Oral Hygiene
MeSH Terms: conditions — Dental Caries | interventions — Clove Oil

STUDY DESIGN:
Intervention Model Description: This study uses a parallel group randomized controlled trial design with three intervention arms: coconut oil pulling with clove oil, coconut oil pulling alone, and fluoride mouthwash (control). The study evaluates the impact on Streptococcus mutans count in children.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study will implement triple blinding, where the participants, investigator, and outcome assessors will be unaware of group allocations to reduce bias in results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: → Coconut Oil Pulling with Clove Oil (Experimental): Arm 1: Coconut Oil Pulling with Clove Oil
  Arm Description:
  Participants in this group will swish 10 mL of coconut oil mixed with 2 drops of clove oil once daily for 4 weeks. The aim is to evaluate its effect on reducing Streptococcus mutans levels in children.
  Interventions: Behavioral: coconut oil pulling with clove oil
- Arm 2: → Coconut Oil Pulling (Experimental): Arm 2: Coconut Oil Pulling
  Arm Description:
  Participants in this group will swish 10 mL of pure coconut oil once daily for 4 weeks. This arm assesses the impact of coconut oil alone on Streptococcus mutans reduction in children.
  Interventions: Behavioral: coconut oil pulling
- Arm 3: → Fluoride Mouthwash (Active Comparator): Arm 2: Coconut Oil Pulling
  Arm Description:
  Participants in this group will swish 10 mL of pure coconut oil once daily for 4 weeks. This arm assesses the impact of coconut oil alone on Streptococcus mutans reduction in children.
  Interventions: Drug: Fluoride Mouthwash

INTERVENTIONS:
Behavioral: coconut oil pulling with clove oil — Participants will swish 10 mL of coconut oil mixed with 2 drops of clove oil once daily for 4 weeks. This intervention is designed to assess its antimicrobial efficacy in reducing Streptococcus mutans levels in children and improving oral hygiene.
  Arms: Arm 1: → Coconut Oil Pulling with Clove Oil
Behavioral: coconut oil pulling — Participants will swish 10 mL of pure coconut oil once daily for 4 weeks. This intervention aims to evaluate the effectiveness of coconut oil alone in reducing Streptococcus mutans levels and its potential role in maintaining oral health.
  Arms: Arm 2: → Coconut Oil Pulling
Drug: Fluoride Mouthwash — Participants will rinse with 10 mL of fluoride mouthwash three times daily for 4 weeks. This intervention serves as the active comparator, as fluoride mouthwash is a well-established method for reducing Streptococcus mutans levels and preventing dental caries.
  Arms: Arm 3: → Fluoride Mouthwash

SUMMARY:
This study aims to compare the effectiveness of coconut oil pulling with clove oil, coconut oil pulling alone, and fluoride mouthwash in reducing Streptococcus mutans levels in children aged 6-12 years. Participants will be randomly assigned to one of three groups:

1. Coconut Oil Pulling with Clove Oil Group - Daily swishing with coconut oil mixed with clove oil.
2. Coconut Oil Pulling Group - Daily swishing with coconut oil alone.
3. Fluoride Mouthwash Group (Control) - Using fluoride mouthwash as per standard guidelines.

The primary outcome is the reduction in Streptococcus mutans count, assessed through microbiological analysis of saliva samples at baseline, immediately after intervention, and after 4 weeks. Secondary outcomes include patient acceptability, adherence, and gingival health.

This randomized controlled trial will provide insight into natural alternatives for oral health maintenance in children.

Study Location: Cairo University, Faculty of Dentistry. Estimated Study Duration: May 2025 - January 2026.

DETAILED DESCRIPTION:
This study is a three-arm, randomized controlled trial assessing the impact of coconut oil pulling with clove oil compared to coconut oil alone and fluoride mouthwash on Streptococcus mutans reduction in children. Participants will be recruited from the Pediatric Dentistry Department at Cairo University and randomly assigned using a 1:1:1 allocation ratio.

Saliva samples will be collected at three time points (baseline, immediately after intervention, and 4 weeks post-intervention) for microbiological analysis. The study will also evaluate secondary outcomes such as patient compliance (measured using the MMAS-4 scale), acceptability (using a 5-point Likert scale), and gingival health (assessed with the Löe & Silness Gingival Index).

The findings aim to determine whether natural oil-based methods can serve as effective, non-invasive alternatives to fluoride-based mouth rinses in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* 1.Children aged 6-12 years old. 2.Both male and female participants. 3.Patients in good general health condition with no systemic disease. 4.Patients' first guardians must provide written informed consent to participate in the study

Exclusion Criteria:

* 1.Patients who have recently received fluoride treatments (within the last 2 weeks).

  2.Patients with a history of recent antibiotic administration (within the last 2 weeks).

  3.Patients who have recently used antimicrobial mouth rinses in the last 12 hours or topical fluoride treatments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
streptococcus mutans count | Baseline (T0), immediately after intervention (T1), and after 4 weeks (T2).
  The primary outcome of this study is the reduction in Streptococcus mutans count in plaque samples collected from participants. Samples will be collected at three time points: baseline (T0), immediately after the intervention (T1), and four weeks post-intervention (T2). The bacterial count will be analyzed using Mitis Salivarius Bacitracin (MSB) Agar and expressed as colony-forming units per milliliter (CFU/mL). The count will be manually determined using a colony counter after incubation under anaerobic conditions for 24-72 hours at 37°C. Gram staining, catalase test, and sugar fermentation tests will be performed to confirm the presence of Streptococcus mutans

CONTACTS AND LOCATIONS:
Overall Officials: nada wassef main supervisor, associate professor, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry-Cairo university, Cairo, Cairo Governorate
  - Faculty of Dentistry Cairo university, Egypt, Cairo Governorate

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional and ethical considerations.